CLINICAL TRIAL: NCT02091167
Title: Prefrontal Modulation by Repetitive Bilateral Transcranial Direct Current Stimulation (tDCS) in Crack-cocaine Addicted Inpatients.
Brief Title: Bilateral Prefrontal Modulation in Crack-cocaine Addiction
Acronym: tDCS_CRACK
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Federal University of Espirito Santo (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Harvard Medical School (HMS and HSDM) (Other); University of Göttingen (Other)
Responsible Party: Principal Investigator, Ester Miyuki Nakamura-Palacios, MD, PhD, Federal University of Espirito Santo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: tDCS CRACK CEP_UFES 384281; CNPq_ 475232/2013-5 (Other Grant/Funding Number: CNPq process # 475232/2013-5)
Record Dates: First submitted 2014-03-16; First posted 2014-03-19 (Estimated); Results first posted 2019-06-24 (Actual); Last update posted 2019-06-24 (Actual); Status verified 2019-03

CONDITIONS: Drug Addiction; Executive Dysfunction
Keywords: crack-cocaine addiction; tDCS; dlPFC; craving; cognition
MeSH Terms: conditions — Substance-Related Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Sham-controlled double-blind randomized clinical trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- real tDCS (Experimental): Ten sessions (every other day) of bilateral transcranial Direct Current Stimulation (tDCS: 2 milliamperes, 3 x 7 cm2, during 20 minutes) over dorsolateral Prefrontal Cortex (cathodal left / anodal right).
  Interventions: Device: transcranial Direct Current Stimulation
- sham-tDCS (Sham Comparator): Ten sessions (every other day) of placebo control (sham procedure) of transcranial Direct Current Stimulation (sham-tDCS) during 20 minutes with electrodes placed over the dorsolateral Prefrontal Cortex (cathodal left / anodal right). Current was delivered for 30 seconds and was turned off for the rest of the stimulation period. In this way, subjects experienced the initial itching sensation at the beginning of stimulation, but received no current for the rest of the session.
  Interventions: Device: transcranial Direct Current Stimulation

INTERVENTIONS:
Device: transcranial Direct Current Stimulation — Direct currents are transferred via a pair of carbonated-silicone electrodes (35 cm2) with a thick layer of high conductive gel for EEG underneath them. The electric current is delivered by an electric stimulator. To stimulate the left DLPFC, the cathode electrode is placed over F3 according to the 10-20 international system while the anode is placed over the contralateral F4 region. The currents flows continuously for 20 minutes with an intensity of 2 milliamperes.
  Other Names: tDCS

SUMMARY:
In this study, eligible crack-cocaine addicted inpatients recruited from specialized clinics for substance abuse disorder treatment, filling inclusion criteria and not showing any exclusion criteria, were randomized to receive the repetitive (10 sessions, every other day) bilateral dorsolateral Prefrontal Cortex (dlPFC: cathodal left / anodal right) tDCS (2 milliamperes, 3x7 cm2, for 20 min) or placebo (sham-tDCS). Craving to the use of crack-cocaine was examined before (baseline), during and after the end of the tDCS treatment.

Based in our previous data, our hypothesis was that repetitive bilateral tDCS over dlPFC would favorably change clinical, cognitive and brain function in crack-cocaine addiction and these would be long-lasting effects.

DETAILED DESCRIPTION:
Before (baseline) and after tDCS or sham-tDCS treatment, subjects were examined:

(1) clinically, regarding craving (obsessive compulsive scale) and relapses to the drug use.

They were followed-up for clinical examination at least 60 days after treatment.

ELIGIBILITY:
Inclusion Criteria:

* patients between the age of 18 and 60 years;
* met criteria for crack-cocaine dependence according to the Diagnostic and Statistical Manual of Mental Disorders, fifth edition (DSM-5), as determined by clinical evaluation;
* in stable clinical condition with no need for inpatient care;
* able to read, write, and speak Portuguese; and
* no severe withdrawal signs or symptoms at baseline.

Exclusion Criteria:

* a condition of intoxication or withdrawal due to a substance other than crack-cocaine;
* unstable mental or medical disorder or substance abuse or addiction other than crack-cocaine dependence, except nicotine and/or caffeine;
* a diagnosis of epilepsy, convulsions;
* a previous history of drug hypersensitivity or adverse reactions to diazepam or other benzodiazepines and haloperidol;
* any contraindication for electrical brain stimulation procedures such as electronic implants or metal implants;
* suspected pregnancy for female participants;

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ester MN Palacios, MD, PhD, Study Director — Federal University of Espírito Santo
Locations (1):
- Federal University of Espírito Santo, Vitória, ES - Espírito Santo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Conti CL, Nakamura-Palacios EM. Bilateral transcranial direct current stimulation over dorsolateral prefrontal cortex changes the drug-cued reactivity in the anterior cingulate cortex of crack-cocaine addicts. Brain Stimul. 2014 Jan-Feb;7(1):130-2. doi: 10.1016/j.brs.2013.09.007. Epub 2013 Oct 12. PMID 24139147
- [Background] da Silva MC, Conti CL, Klauss J, Alves LG, do Nascimento Cavalcante HM, Fregni F, Nitsche MA, Nakamura-Palacios EM. Behavioral effects of transcranial direct current stimulation (tDCS) induced dorsolateral prefrontal cortex plasticity in alcohol dependence. J Physiol Paris. 2013 Dec;107(6):493-502. doi: 10.1016/j.jphysparis.2013.07.003. Epub 2013 Jul 25. PMID 23891741
- [Background] Nakamura-Palacios EM, Souza RS, Zago-Gomes MP, de Melo AM, Braga FS, Kubo TT, Gasparetto EL. Gray matter volume in left rostral middle frontal and left cerebellar cortices predicts frontal executive performance in alcoholic subjects. Alcohol Clin Exp Res. 2014 Apr;38(4):1126-33. doi: 10.1111/acer.12308. Epub 2013 Nov 20. PMID 24256621
- [Background] de Souza Custodio JC, Martins CW, Lugon MD, Fregni F, Nakamura-Palacios EM. Epidural direct current stimulation over the left medial prefrontal cortex facilitates spatial working memory performance in rats. Brain Stimul. 2013 May;6(3):261-9. doi: 10.1016/j.brs.2012.07.004. Epub 2012 Aug 1. PMID 22878259
- [Background] Batista EK, Klauss J, Fregni F, Nitsche MA, Nakamura-Palacios EM. A Randomized Placebo-Controlled Trial of Targeted Prefrontal Cortex Modulation with Bilateral tDCS in Patients with Crack-Cocaine Dependence. Int J Neuropsychopharmacol. 2015 Jun 10;18(12):pyv066. doi: 10.1093/ijnp/pyv066. PMID 26065432
- [Background] Nakamura-Palacios EM, Lopes IB, Souza RA, Klauss J, Batista EK, Conti CL, Moscon JA, de Souza RS. Ventral medial prefrontal cortex (vmPFC) as a target of the dorsolateral prefrontal modulation by transcranial direct current stimulation (tDCS) in drug addiction. J Neural Transm (Vienna). 2016 Oct;123(10):1179-94. doi: 10.1007/s00702-016-1559-9. Epub 2016 Apr 30. PMID 27138429
- [Background] Klauss J, Anders QS, Felippe LV, Nitsche MA, Nakamura-Palacios EM. Multiple Sessions of Transcranial Direct Current Stimulation (tDCS) Reduced Craving and Relapses for Alcohol Use: A Randomized Placebo-Controlled Trial in Alcohol Use Disorder. Front Pharmacol. 2018 Jul 3;9:716. doi: 10.3389/fphar.2018.00716. eCollection 2018. PMID 30018558
- [Background] de Souza Custodio JC, Martins CW, Lugon MDMV, de Melo Rodrigues LC, de Figueiredo SG, Nakamura-Palacios EM. Prefrontal BDNF Levels After Anodal Epidural Direct Current Stimulation in Rats. Front Pharmacol. 2018 Jul 12;9:755. doi: 10.3389/fphar.2018.00755. eCollection 2018. PMID 30050442
- [Background] Klauss J, Penido Pinheiro LC, Silva Merlo BL, de Almeida Correia Santos G, Fregni F, Nitsche MA, Miyuki Nakamura-Palacios E. A randomized controlled trial of targeted prefrontal cortex modulation with tDCS in patients with alcohol dependence. Int J Neuropsychopharmacol. 2014 Nov;17(11):1793-803. doi: 10.1017/S1461145714000984. Epub 2014 Jul 10. PMID 25008145
- [Background] Anders QS, Klauss J, Rodrigues LCM, Nakamura-Palacios EM. FosB mRNA Expression in Peripheral Blood Lymphocytes in Drug Addicted Patients. Front Pharmacol. 2018 Oct 24;9:1205. doi: 10.3389/fphar.2018.01205. eCollection 2018. PMID 30405417
- [Background] Martins CW, de Melo Rodrigues LC, Nitsche MA, Nakamura-Palacios EM. AMPA receptors are involved in prefrontal direct current stimulation effects on long-term working memory and GAP-43 expression. Behav Brain Res. 2019 Apr 19;362:208-212. doi: 10.1016/j.bbr.2019.01.023. Epub 2019 Jan 14. PMID 30654123
- [Result] Klauss J, Anders QS, Felippe LV, Ferreira LVB, Cruz MA, Nitsche MA, Nakamura-Palacios EM. Lack of Effects of Extended Sessions of Transcranial Direct Current Stimulation (tDCS) Over Dorsolateral Prefrontal Cortex on Craving and Relapses in Crack-Cocaine Users. Front Pharmacol. 2018 Oct 23;9:1198. doi: 10.3389/fphar.2018.01198. eCollection 2018. PMID 30405414

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were two dropouts in the sham-tDCS group that were excluded after randomization. One patient escaped from the treatment facility and the other had to be discontinued because of precocious discharge from the clinic for misconduct.
Period: Overall Study
Arm/Group | Real tDCS | Sham-tDCS
Started | 19 | 16
Completed | 19 | 14
Not Completed | 0 | 2
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Real tDCS | Sham-tDCS | Total
Number analyzed (Participants) | 19 | 14 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.1 (9.6) | 35.0 (8.2) | 35.03 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 15 | 12 | 27
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Years of education [Count of Participants; unit: Participants]
  Between 6 to 9 | 7 | 4 | 11
  Between 10 to 13 | 8 | 7 | 15
  Above 13 | 4 | 3 | 7
Employment situation [Count of Participants; unit: Participants]
  Formal job | 2 | 4 | 6
  Unemployed | 9 | 8 | 17
  Freelance | 7 | 1 | 8
  Retired | 1 | 1 | 2
Marital state [Count of Participants; unit: Participants]
  Single | 12 | 10 | 22
  Married | 2 | 0 | 2
  Common-law | 0 | 1 | 1
  Divorced | 1 | 2 | 3
  Widow | 0 | 1 | 1
  Non reported | 4 | 0 | 4
Tobacco use [Count of Participants; unit: Participants]
  Yes | 11 | 11 | 22
  No | 8 | 3 | 11

OUTCOME MEASURES:

1. Primary Outcome: Craving
Description: Five items from the original obsessive compulsive drinking scale, which are believed to reliably assess craving in a narrow sense were used. Questions of this brief scale allow quantification of thoughts and feelings (obsessions), and behavioral intentions, and are answered on a scale ranging from 0 to 4, resulting in a total score between 0 and 20.
  Higher scores reflect more severe craving. These items were applied at the beginning, during and at the end of the treatment with sham-tDCS or tDCS.
Time Frame: Five applications: once in the week before tDCS treatment (baseline), second, third and fourth weeks, during the treatment, and in the fith week, after the end of the tDCS treatment.
Population: Two patients from each group were lost to follow-up after their discharge from the hospital.
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- Real-tDCS: Crack-cocaine patients who underwent 10 sessions of real tDCS treatment.
- Sham-tDCS: Crack-cocaine patients who underwent sham (placebo)-tDCS control procedure.
Arm/Group | Real-tDCS | Sham-tDCS
Number analyzed (Participants) | 19 | 14
scores on a scale
  1 | 6.53 (5.2) | 7.0 (3.8)
  2 | 4.74 (4.1) | 4.43 (2.9)
  3 | 3.63 (3.9) | 4.0 (3.2)
  4 | 2.63 (3.4) | 3.5 (3.1)
  5 | 2.26 (2.9) | 4.07 (3.4)
Statistical Analysis 1: Comparison: Real-tDCS vs Sham-tDCS; We powered for a medium effect size based on our previous study with effect size (partial ղ2) of 0.10384 for the main within-subject factor in the two-way ANOVA with repeated measures. With a power of 80%, and a two-sided probability of a type I error of 5%, the resulting minimum sample size was 30 participants. To account for waiving or dropouts we increased the estimated sample size to approximately 10%, resulting in 33 subjects in total (approximately 16 to 17 subjects in each group); Test type: Other; p = 0.05, ANOVA; Most of data (age, patterns of crack-cocaine use, 5-items OCCS) were normally distributed according to the D'Agostino & Pearson normality test, thus they were analyzed by parametric tests. Between-group (sham- and real tDCS) comparisons were conducted by unpaired Student´s t-tests. For all other non-parametric data (gender, schooling, employment, marital state and tobacco use), Chi-square or Fisher tests were used to compare sham and real tDCS groups. Besides the two-way ANOVA with repeated measures followed by Bonferroni-corrected t-tests, linear regression analyses were done over craving scores obtained along the 4-week treatment (five time-points measurements) for both groups. Additional comparisons between initial and final OCDS scores were done by paired t-tests for each group, and differences between final and initial scores were compared between sham-tDCS and real tDCS groups with unpaired t-test

2. Primary Outcome: Relapses
Description: A use relapse was defined as the first episode of return to the previous uncontrolled pattern of crack-cocaine use (rocks per day). Information about relapse were gathered directly when patients regularly returned to the hospital for clinical follow-up after their discharge and/or by self-report or reports of family members by telephone calls.
Time Frame: 30 and 60 days after discharge from clinics
Measure: Count of Participants; unit: Participants
Arm/Group | Real-tDCS | Sham-tDCS
Number analyzed (Participants) | 17 | 12
Participants
  30-days follow-up: Not relapsed | 10 | 7
  30-days follow-up: Relapsed | 7 | 5
  60-days follow-up: Not relapsed | 8 | 4
  60-days follow-up: Relapsed | 9 | 8
Statistical Analysis 1: Comparison: Real-tDCS vs Sham-tDCS; Two patients from each group were lost to follow-up after their discharge from the hospital; Test type: Other; p = 0.05, Fisher Exact

ADVERSE EVENTS:
Time Frame: Adverse events were examined once at the end of each tDCS application. Therefore, over 10 tDCS applications, with a total of 10 examinations.
Description: We asked subjects about the following adverse effects: headache, neck and scalp pain, tingling, itching, skin redness, burning sensation of the scalp, sleepiness, acute mood changes, trouble concentrating, and others after treatment.
Arm/Group | Real-tDCS | Sham-tDCS
All-Cause Mortality (participants affected / at risk) | 0/19 | 2/14
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/14
Other Adverse Events (participants affected / at risk) | 16/19 | 8/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Real-tDCS (N=19) | Sham-tDCS (N=14)
Tingling in the scalp (Skin and subcutaneous tissue disorders) | 14 (14) | 7 (7)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Drowsiness (Nervous system disorders) | 1 (1) | 0 (0)
Burning sensation of the scalp (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Sample size restricted by inclusion and exclusion criteria, limiting generalizability of our results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-23): https://cdn.clinicaltrials.gov/large-docs/67/NCT02091167/Prot_SAP_000.pdf